CLINICAL TRIAL: NCT05102435
Title: Cross-cultural Translation and Validation of the Performance Oriented Mobility Assessment (Poma) Scale Into Urdu Version
Brief Title: Translation and Validation of the Performance Oriented Mobility Assessment (Poma) Scale Into Urdu Version
Status: Completed | Type: Observational
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Other Study IDs: REC/00964 Kiran
Record Dates: First submitted 2021-10-19; First posted 2021-11-01 (Actual); Last update posted 2022-04-29 (Actual); Status verified 2022-04

CONDITIONS: Fall

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Tool Translation & Validation study — In this English version of POMA scale will be translated into Urdu.

SUMMARY:
The aim of this study is to translate the original English version POMA scale into Urdu and also determine cultural adaptation to establish its validity and reliability. This study also aims to correlate Performance oriented Mobility Assessment (POMA) scales with time up and go test in elderly population.

DETAILED DESCRIPTION:
Among older persons, age-related impairments cause loss of postural control and balance that result in pain, independency and disability. One of the most common geriatric syndromes and most serious health issue threatening the independency of older persons is fall. The impact of these fall-related injuries on older person, families and societies and its fruitful intervention has made this issue important worldwide. Approximately 28-35% of people aged 65 years and 32-42% of aged 70 years' experience falls annually and 10% suffer serious injury such as, fracture, severe head trauma and joint dislocation. The incidence rate of fall is higher in hospitalized and residents of nursing home. It rises from middle age and peaks in person above 80 years. The risk factors associated with falls are, lower extremity muscle weakness, gait or balance deficits, use of an assistive device, cognitive impairment, visual deficit, arthritis and impaired activities of daily living . Different scales and tests are used for risk factors for falls, balance and mobility such as Berg Balance Scale, Time up and go test and dynamic gait index and Fullerton Advanced Balance Scale. One of these scales Performance-Oriented Mobility Assessment (POMA) scale. POMA scale has acceptable reliability and validity as compared to FRT and TUG in elderly. The advantages of this scale are; applicability, low cost, easy to administer, no equipment is needed other than a standard chair and stopwatch, evaluates functional activities and assesses both balance (POMA-B) and gait components (POMA-G)Originally POMA scale was used to assess risk of fall in institutionalized populations but later on used as an assessment tool for mobility and determine effects of interventions.

The POMA has found to be widely used in patients who have dynamic and reactive balance deficits. It comprises 16 items (9 balance and 7 gait related). Total time taken for administration is approximately 10 minutes and total score is 28; 16 is balance and 12 is gait score. Some Items are scored dichotomously (can/cannot perform) and others are scored 0, 1 or 2 points for quality of performance. The higher scores show low fall risk and better balance while lower score predicts poorer balance and greater risk of fall. The score 19-24/28 indicates moderate risk for falling while score <19 indicates a "high" risk for falling.

ELIGIBILITY:
Inclusion Criteria:

* The sample will be assessed a cognition evaluation through the mini-mental test
* Any present or previous history of vertigo since last 6 months

Exclusion Criteria:

* Patients with any neurological disorder,
* previous orthopedic surgery within last 6 months,
* bedridden,
* wearing any prosthesis, and illiteracy.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Performance-oriented Mobility Assessment (POMA) is one of the functional measures used to evaluate balance, gait, and fall risk in the elderly.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-03-31 (Actual)

PRIMARY OUTCOMES:
Performance oriented mobility Assessment scale | 1 time assessment of mobility and balance (approximately 10 minutes)
  Performance oriented mobility Assessment scale is used to assess risk of fall in institutionalized populations but later on used as an assessment tool for mobility and balance assessment. Total time taken for administration is approximately 10 minutes and total score is 28; 16 is balance and 12 is gait score

CONTACTS AND LOCATIONS:
Overall Officials: Misbah ghous, MS, Principal Investigator — Riphah International University Islamabad
Locations (1):
- Misbah Ghous, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Yücel SD, Şahin F, Doğu B, Şahin T, Kuran B, Gürsakal S. Reliability and validity of the Turkish version of the Performance-Oriented Mobility Assessment I. European Review of Aging and Physical Activity. 2012 Oct;9(2):149-59.
- [Background] Schulein S, Pflugrad L, Petersen H, Lutz M, Volland-Schussel K, Gassmann KG. [German translation of the performance-oriented mobility assessment according to Tinetti]. Z Gerontol Geriatr. 2017 Aug;50(6):498-505. doi: 10.1007/s00391-016-1070-9. Epub 2016 Jun 16. German. PMID 27312196
- [Background] Moulodi B, Azad A, Taghizadeh G, Roohi-Azizi M, Mohammadi P. Reliability and validity of persian version of performance-oriented mobility assessment (POMA) in Community-dwelling Iranian Older Adults: Psychometric Properties. Iranian Rehabilitation Journal. 2020;18(1):39-48.